CLINICAL TRIAL: NCT01162304
Title: Open-Label Trial Comparing Oxycodone Medications for Effectiveness and Satisfaction (OUTCOMES)
Brief Title: Open-Label Trial Comparing Oxycodone Medications
Acronym: OUTCOMES
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: unable to enroll subjects meeting Eligibility criteria
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Joel Kent, Principal investigator, University of Rochester
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 29813
Record Dates: First submitted 2010-04-27; First posted 2010-07-14 (Estimated); Results first posted 2015-07-17 (Estimated); Last update posted 2015-07-17 (Estimated); Status verified 2014-01

CONDITIONS: Chronic Pain
Keywords: Chronic Pain; This clinical trial will compare immediate-release (IR); oxycodone and extended-release (ER) oxycodone in the; management of chronic pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ER Oxycodone vs IR Oxycodone (Active Comparator): Extended release Oxycodone to assess pain relief adverse effects, treatment satisfaction and impact of treatment on health related quality of life.
  IR oxycodone will be distributed to subjects in 5 mg pills and they will be instructed to take 3-4 of these pills every four hours
  Interventions: Drug: Extended Release Oxycodone; Drug: Immediate Release Oxycodone

INTERVENTIONS:
Drug: Extended Release Oxycodone — 40 mg tablets one to two every 12 hours, Immediate release 5mg pills 1-2 tablets every 6 hours
  Other Names: Medication comparison
Drug: Immediate Release Oxycodone — IR oxycodone will be distributed to subjects in 5 mg pills and they will be instructed to take 3-4 of these pills every 4 hours
  Other Names: Medication comparison

SUMMARY:
The investigators hypothesize that subjects will have greater pain relief when taking IR-oxycodone compared with ER-oxycodone for several reasons. The ability to take a varying amount of medication at six different points over the course of a day will allow patients to take as much (or as little) medication as they need to control their pain. In addition, the ability to vary the medication doses in this way will give them a greater sense of control, which will also contribute to greater pain relief. Similarly, the investigators predict that patients will show greater benefits with IR-oxycodone on the measures of physical and emotional functioning. Because there is relatively little data on sleep apnea in chronic pain patients (Webster et al., 2008), these assessments are exploratory and not hypothesis-based. Finally, although it is typically thought that the abuse liability of IR-opioid medications is greater than for ER-medications, the data on which this belief are based have not involved systematic studies of patients with chronic pain; the assessments of abuse liability will therefore also be exploratory.

DETAILED DESCRIPTION:
This study is a single-center, randomized, open-label, 13-week, 2-period crossover clinical trial. Subjects will complete each of the following (unless they withdraw from the trial): (1) a one-week baseline period during which the subject completes pain diaries and remains on stable dosages of their existing pain medications; (2) immediate-release (IR) oxycodone 5 mg 3-4 pills every four hours; (3) extended-release (ER) oxycodone 40 mg 1 pill every 12 hours and IR-oxycodone 5 mg 1-2 pills every six hours. Subjects will be randomized to one of two treatment sequences (ER-oxycodone first then IR-oxycodone or vice verse). It is expected that this trial will take approximately 2 years to complete.

Crossover periods. Each of the two treatment periods will be 6 weeks in duration, which will allow ample time to assess pain relief, adverse effects, treatment satisfaction, and impact of treatment on health-related quality of life. There will be no need for a titration period at the beginning of either period or for a washout period before the second period because oxycodone at the same dosages will be administered in both periods. At each visit, subjects will be given sufficient medication to sustain them until at least the following visit.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 18 years old.
2. Be able to read and understand English.
3. Have a diagnosed chronic pain condition with pain every day or most days for the previous 6 months.
4. Be receiving the equivalent of no more than 40-120 mg daily of an opioid analgesic that can be safely converted to oxycodone; this dosage includes all use of opioid analgesics, including for "rescue" and for "breakthrough" pain.
5. Have an average daily pain rating for the baseline week of pain ratings equal to 4.0 or greater on a 0-10 numerical pain rating scale (NRS) of average pain intensity in the past 24 hours.
6. Have completed at least 6 of the 7 daily diaries during the baseline week.
7. Have at least 5 baseline week pain diary ratings equal to 3 or greater on the 0-10 NRS, with no more than one rating of 9 and no ratings of 10.
8. Have stable concomitant use of all pain-related medications for 8 weeks prior to screening and being willing to continue stable use of these medications for the duration of the trial.
9. Have the ability to either independently or with an accompanying person come to the research center for study visits.

Exclusion Criteria:

1. Treatment of their chronic pain with nerve blocks or any other interventional procedure within the past 8 weeks.
2. A Beck Depression Inventory score < 27 at baseline or clinically significant depression or dementia that, in the opinion of the investigator, may interfere with a subjects' adherence to the study protocol and/or the accurate and consistent reporting of pain.
3. History of suicide attempt within the past 2 years or current suicide plan or intent.
4. History of excessive alcohol use or any illicit drug use within the past 2 years.
5. Lack of adequate birth control in pre-menopausal women of child-bearing age and/or a positive urine pregnancy test, which will be performed on all women except those > 2 years post-menopausal or who have had a hysterectomy).
6. History of malignancy within the past five years with the exception of successfully treated non-metastatic basal cell or squamous cell carcinomas of the skin.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel L Kent, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1-20-2010 to 11-21-2013 at the medical center.
Pre-assignment Details: Study was terminated participants were enrolled but treatment arm assigment was not shared with the study team.The study team was blinded and research pharmacy which was tracking randomization destroyed study records before sharing with the study team.
Groups:
- ER Oxycodone vs IR Oxycodone: Extended release Oxycodone to assess pain relief adverse effects, treatment satisfaction and impact of treatment on health related quality of life.
  Extended Release Oxycodone: 40 mg tablets one to two every 12 hours, Immediate release 5mg pills 1-2 tablets every 6 hours
  IR oxycodone will be distributed to subjects in 5 mg pills and they will be instructed to take 3-4 of these pills every four hours Immediate Release Oxycodone: IR oxycodone will be distributed to subjects in 5 mg pills and they will be instructed to take 3-4 of these pills every 4 hours
Period: Overall Study
Arm/Group | ER Oxycodone vs IR Oxycodone
Started | 18
Completed | 7
Not Completed | 11
Not completed — Beck scale to high | 11

BASELINE CHARACTERISTICS:
Arm/Group | ER Oxycodone vs IR Oxycodone
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 9
  More than one race | 0
  Unknown or Not Reported | 7
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Numerical Pain Rating Scale (NRS)
Description: The primary outcome measure for this clinical trial will be pain relief documented in the subjects' daily pain diaries. Specifically, the average of the daily pain ratings recorded by subjects during the final weeks of the two treatment periods will be compared. The treatment comparison of interest is IR-oxycodone vs. ER-oxycodone, which will be tested at the p < 0.05 level using a two-tailed test.
Time Frame: Daily
Population: Due to not reaching enrollment goal of 40 subjects, data collected on the 7 participants enrolled was not analyized because the data is not available the data are locked not able to obtain.
Groups:
- Extended Release Oxycodone: Extended release Oxycodone to assess pain relief adverse effects, treatment satisfaction and impact of treatment on health related quality of life.
  Extended Release Oxycodone: 40 mg tablets one to two every 12 hours, Immediate release 5mg pills 1-2 tablets every 6 hours
- Immediate Release Oxycodone: IR oxycodone will be distributed to subjects in 5 mg pills and they will be instructed to take 3-4 of these pills every four hours
  Immediate Release Oxycodone: IR oxycodone will be distributed to subjects in 5 mg pills and they will be instructed to take 3-4 of these pills every 4 hours
Arm/Group | Extended Release Oxycodone | Immediate Release Oxycodone
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Brief Pain Inventory
Description: Will be administered to assess the extent to which chronic pain interferes with sleep and physical and emotional functioning.
Time Frame: Visits 2-6
Population: as for outcome 1
Arm/Group | Extended Release Oxycodone | Immediate Release Oxycodone
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Hospital Anxiety and Depression Scale
Description: The HADS will be administered to assess anxiety and depression.
Time Frame: Visits 2-6
Population: as for outcome 1
Arm/Group | Extended Release Oxycodone | Immediate Release Oxycodone
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Short Form Health Survey (SF-36)
Description: It is a 36-item questionnaire designed to measure general health related quality of life.
Time Frame: Visits 2, 4 and 6
Population: as for outcome 1
Arm/Group | Extended Release Oxycodone | Immediate Release Oxycodone
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Patient Global Impression of Change
Description: This rating on a 7-point scale measures a patients overall assessment of change since starting a given treatment. This measure provides a subjects global assessment of change, presumably including change in pain, side effects, change in functional status, convenience of therapy, subject preference and values and overall satisfaction with the intervention.
Time Frame: Visits 4 and 6 the end of each of the two treatment periods
Population: as for outcome 1
Arm/Group | Extended Release Oxycodone | Immediate Release Oxycodone
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Extended Release Oxycodone | Immediate Release Oxycodone
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes